CLINICAL TRIAL: NCT07240220
Title: The Mother-Daughter Project: Inclusion of Difficult-to-reach Kenyan Families, and Studies of Factors Influencing the Immune Response to HPV Vaccination (Merck-4)
Brief Title: The Mother-Daughter Project: Merck-4
Acronym: Merck-4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Darron Brown MD, MPH, Professor of Microbiology, Indiana University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Merck-4 (irb 28570) (102790); 102790 (Other: Merck)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Cervical Dysplasia
Keywords: cervical dysplasia; cervical cancer screening; HPV infection
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections | interventions — Watchful Waiting; Acetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kenyan women (Other): Up to 500 adult women will undergo cervical cancer screening.
  Interventions: Diagnostic Test: High Risk HPV DNA Testing; Procedure: Visual Inspection with acetic acid (VIA) and possible cervical biopsy
- Kenyan daughters (Other): Up to an additional 2000 girls (daughters of participants in the Kenyan women arm) will be immunized against HPV using the 9-valent HPV vaccine (Gardasil-9).
  Interventions: Biological: Gardisil-9

INTERVENTIONS:
Biological: Gardisil-9 — The 9 valent vaccine will be offfered to 2000 adolescent girls. The 9 valent vaccine will be offered to 2000 adolescent girls. The first vaccination dose will be administered at a community meeting, after parental consent has been obtained. The second vaccination dose will be administered at a subsequent community meeting, 6 to 12 months after the first dose.
  Other Names: 9-valent HPV vaccine
  Arms: Kenyan daughters
Diagnostic Test: High Risk HPV DNA Testing — Self-collected cervical swabs will be tested for high-risk HPV using the Roche Cobas Assay. This assay provides specific HPV 16 or 18 detection, as well as detection of any of 12 additional oncogenic types (HPV types 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68).
  Arms: Kenyan women
Procedure: Visual Inspection with acetic acid (VIA) and possible cervical biopsy — Cervical screening in Kenya is usually done through pelvic examination and VIA. Cervical biopsy will additionally be performed for all HIV-infected women, and for HIV-uninfected women with abnormal VIA results.
  Arms: Kenyan women

SUMMARY:
This project serves to continue a community-based initiative, known as the Kenya Mother-Daughter Cervical Cancer Eradication Project, or the Mother-Daughter Project (MDP), in the Webuye region of Western Kenya. The MDP project, since its initiation in 2018, has sought to develop a framework for the eradication of cervical cancer through effective screening of adult women and through the vaccination of female children.

This project specifically aims to collect additional data on the ability for HR-HPV testing to detect premalignant lesions of the cervix, especially in HIV-infected women, to investigate and identify barriers leading to non-participation in previous MDP efforts, and to examine factors associated with the immune response to HPV vaccination among rural Kenyan girls.

DETAILED DESCRIPTION:
Cervical cancer is caused by oncogenic, or "high-risk" (HR) human papillomavirus (HPV) and is the main cause of cancer-related death among Kenyan women. Although preventable, this malignancy occurs frequently in women living in rural areas of Kenya where screening is seldom performed, and girls are not vaccinated against HPV. Only 5% of Kenyan women are regularly screened, and 14% have ever been screened, done in Kenya by a method known as Visual Inspection with Acetic Acid (VIA). Obstacles to effective screening include long travel to clinics, high costs, and factors related to VIA such as poor sensitivity and specificity, the need for practitioner training for VIA, variability among providers in VIA interpretation, and others. In addition, while safe and effective HPV vaccines have been available since 2006, very few (<5%) Kenyan girls have been vaccinated. Obstacles to vaccination include high costs, poor delivery infrastructure, lack of education, long travel to clinics, and others. Additionally, strategies based on centralized care have been unsuccessful in preventing cervical cancer in Kenyan women.

In 2018, an initiative known as the Kenya Mother-Daughter Cervical Cancer Eradication Project, or the Mother-Daughter Project (MDP), was developed in the Webuye region of Western Kenya. Early work from the MDP demonstrated that self-collection of cervical swabs, and the administration of HPV vaccination, is acceptable and feasible within a community rural setting. This continuation project will further study the utility of this strategy, elucidate the barriers to participation, and begin to provide information about the impact of the program.

An additional cohort of 500 adult women will be enrolled in the cervical cancer screening initiative to strengthen the power of analysis on HR-HPV testing to detect premalignant lesions of the cervix, especially in HIV-infected women (Aim 1). Second, families who were invited to the MDP but declined to participate will be identified to investigate and identify barriers leading to their non-participation of the MDP (Aim 2). Third, vaccination efforts will be expanded through the enrollment of an additional 2000 girls, and factors associated with the immune response to HPV vaccination among 9- to 14-year-old rural Kenyan girls will be examined (Aim 3).

This prospective cohort study will be conducted in Webuye, a community located in the western region of Kenya, in Bungoma County on the highway to Uganda. A "Community Entry Strategy" was utilized to introduce prior studies and to invite women to community meetings. A female Kenyan Counselor was trained about cervical cancer (including the cause and the ways to prevent the cancer), how to educate women about this malignancy and how to instruct women in performance of self-collected swabs. Village chiefs, village elders, women deemed to be community leaders, and leaders of the local churches have been approached by the Counselor and Study Coordinator to discuss the goals, strategy, and risks and benefits of the study; this process will be repeated before the current study is initiated. Discussions have focused on the importance of early screening for cervical cancer, the use of self-collected swabs for screening, and the importance of vaccination of children against HPV.

For Aim 1, an additional 500 Kenyan women between the ages of 25 to 49 years (the government-recommended age range for screening in Kenya) will be enrolled. Only women who did not participate in our MDP studies will be enrolled. Women will be instructed in collecting vaginal swabs during the community meetings, and these self-collected swabs will be given to the Counselor. Swabs will be tested for HR-HPV DNA at Lancet Laboratories in Nairobi (or at Moi University if reagents can be obtained) using the Roche Cobas Assay. All women will be asked to travel to the Webuye Clinic for pelvic examination and VIA (the Kenyan standard of care). Cervical biopsy will be performed on all HIV-infected women and on those HIV-uninfected women with abnormal VIA examinations. Results will be analyzed to determine the sensitivity, specificity, positive predictive value, and negative predictive value for HR-HPV DNA to predict biopsy-proven cervical intraepithelial lesion grades 2 and 3, or invasive cancer (CIN2/3) in the HIV-infected group of women.

For Aim 2, adult women and their daughters (if they have daughters), will be asked to fill out questionnaires that will provide data about educational aspects and overall acceptability of the MDP and obstacles related to its initiation. This will be done following the second vaccine dose that will be administered to girls at community meetings. Women in the Webuye community have been satisfied with self-collection of swabs as a method of cervical cancer screening, and most are willing to have their daughters vaccination against HPV. However, it is important to identify those women who do not want to attend meetings, do not want to provide self-collected swabs, or do not want their daughters vaccinated against HPV infection. These women will be traced through 1) records that will be acquired for all women who attend the community meeting, 2) records about women who refuse to participate, and 3) meeting in person (home visits) with women who decline through their phone contacts, through community leaders who understand their physical locations.

For Aim 3, an additional 2000 girls, ages 9 through 14, will be enrolled and the first 9v HPV vaccine will be administered to these girls at a community meeting. The second dose of the HPV vaccine will be administered six to twelve months after the first dose at a subsequent community meeting. Factors associated with the immunological response to the 9v HPV vaccine will additionally be studied. For that purpose, 120 girls will have a blood sample taken at a community meeting, approximately 24 months after receiving the second 9v HPV vaccine dose. Each girl's BMI will be determined. The blood sample will be analyzed for plasma aflatoxin, antibody titers to each of the nine HPV types represented in the 9v vaccine, and for folate, iron, and hemoglobin. In addition, girls will be interviewed with their mothers regarding specific dietary habits.

ELIGIBILITY:
Kenyan Adult Women

Inclusion Criteria:

* ages 25 through 49 years
* able/willing to sign informed consent
* willing to participate in the community meetings

Exclusion Criteria:

• pregnant

Kenyan Girls

Inclusion Criteria:

* ages 9 through 14 years
* have mother that is able/willing to sign informed consent for vaccination
* can return for the second HPV vaccine dose in 6 - 12 months

Exclusion Criteria:

• girls who are not willing or unable to return for the second HPV vaccine dose

Ages: 9 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Detection of CIN2/3 | Baseline
  Following a community meeting at which education on cervical cancer, self-collection of swabs for analysis and HPV vaccination are discussed, participating adult women will provide a self collected swab that will be analyzed for high risk HPV. All participating adult women will additionally undergo pelvic examination and VIA (the Kenyan standard of care). Cervical biopsy will be performed on all HIV-infected women and those HIV-uninfected women with abnormal VIA examinations.
  For the cohort of women who will undergo cervical biopsy, the rates of HR-HPV positivity, VIA abnormality and CIN2/3 detection will be reported for all women and by HIV status. Sensitivity, specificity, positive predictive value, and negative predictive value between HR-HPV and VIA in the detection of biopsy-proven cervical intraepithelial lesion grades 2 and 3, or invasive cancer (CIN2/3) will be compared.
Local knowledge and attitudes | Baseline and after HPV vaccination of daughters is complete (assessed 2 weeks after second vaccine)
  Adult women and their daughters (if they have daughters), will be asked to fill out questionnaires that will evaluate women's knowledge of cervical cancer screening and HPV vaccination and attitudes towards their own health and health of their daughters.
Barriers to participation | During a one-time interview
  Both women who attend the MDP community meeting but decline to participate, and women in the village who were invited but did not attend the community meeting can be identified by the local counselor. The counselor will later contact these women for an interview to determine the reasons for declining participation. It is expected that 20 non-participants will be interviewed to identify barriers. Specific barriers mentioned by the women will then be grouped into several categories. Potential categories may be "lack of confidence in safety of the procedures" (self-collection swab or HPV vaccination of children), "other obligations competing for time", or "cultural-related inhibition". The frequency and percentage of each specific barrier mentioned by the women will be reported.
Factors that influence immunity to the HPV vaccine | 24 months after second HPV vaccine
  The HPV vaccine will be administered at community meetings to participating girls. Approximately 24 months after receiving the second vaccine dose, a subset of girls will undergo a blood sample and BMI measurement at another community meeting. The blood sample will be analyzed for plasma aflatoxin, for antibody titers to each of the nine HPV types in the vaccine, and for folate, iron, and hemoglobin (indicators of nutrition). The girls will also be interviewed with their mothers regarding specific dietary habits.

CONTACTS AND LOCATIONS:
Locations (1):
- Moi University, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: Undecided